CLINICAL TRIAL: NCT06811649
Title: Comparison of Echo-assisted ALR (Loco-regional Anesthesia) Technique and Traditional ALR Technique for the Placement of an Epidural Catheter in the Obstetric Patient Performed by an Anesthesia Resident
Brief Title: Comparison of Echo-assisted ALR Technique and Traditional ALR Technique for the Placement of an Epidural Catheter in the Obstetric Patient
Acronym: OST-22-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OST-22-01
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy
Keywords: epidural catheter; loco-regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- echo-assisted ALR (loco-regional anesthesia) technique (Experimental): Ultrasound evaluation of the spine as an aid in facilitating the placement of an epidural catheter
  Interventions: Diagnostic Test: Ultrasound guided injection with local anaestethic
- traditional ALR technique (No Intervention): The traditional neuroaxial technique involves palpation of the spinous processes and iliac crests to recognize the median and height of the lumbar interspace to be used to perform a neuroaxial block

INTERVENTIONS:
Diagnostic Test: Ultrasound guided injection with local anaestethic — Experimental treatment consists of ultrasound assessment combined with palpatory assessment to identify the most suitable space for epidural catheter insertion.
  The conventional neuroaxial technique relies on palpation of the spinous processes and iliac crests to recognize the midline and height of the lumbar interspace to be used to perform a neuroaxial block.
  With the echo-assisted technique, in aid of the conventional technique, a preprocedure (Prepuncture) is performed for the purpose of combining classic anatomical findings with useful sonographic findings that should improve the success of the neuroaxial technique.
  Arms: echo-assisted ALR (loco-regional anesthesia) technique

SUMMARY:
This is a randomized, open-label, single-center clinical trial. The purpose of the study is to understand whether the aid of ultrasound assessment is useful in improving the competence of resident.

Specifically, to demonstrate how the aid of echo-assistance in the evaluation of the spine increases the atraumatic success rate (primary objective) and reduces the number of complications (particularly, the number of attempts needed and the rate of dura puncture) (secondary objective) in physicians in specialty training.

Pregnant patients requiring peridural analgesia will be assigned to the intervention or control group by simple randomization.

DETAILED DESCRIPTION:
The use of echo-assisted assessment has been studied for about a decade, showing encouraging results as far as experienced medical personnel are concerned, but to date, a systematic study assessing the usefulness of this aid in improving residents' competence (as indicated by the 2019 systematic review) is lacking in the literature.

To date, echo-assisted assessment is not routinely applied to all obstetric patients, as it is a relatively new technique and not yet widely used by all anesthesiologists.

If the results of the study are positive,echo-assisted assessment use could be expanded, reducing the number of complications and increasing the number of atraumatic epidural catheter placements.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients >18 years of age with no BMI (Body Mass Index) limitation
* Pregnant patients requiring partoanalgesia
* Obtaining informed consent for study participation

Exclusion Criteria:

* Patients with contraindications to epidural catheter placement
* Endocranial hypertension
* Coagulopathies
* Severe thrombocytopenia < 75,000 per mm^3.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant patients
Enrollment: 146 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
the rate of FNP (thus atraumatic puncture) | Through study completion,an average of 1 year
  The primary objective of this study is to demonstrate whether or not the aid of echo-assistance in spinal evaluation, performed by an experienced anesthesiologist, increases the atraumatic success rate, First Needle Pass (FNP), in epidural catheter placement by inexperienced personnel (physicians in specialty training, MFS).
  This objective will be calculated by observing the rate of FNP (thus atraumatic puncture).

SECONDARY OUTCOMES:
Change the number of complications | Through study completion,an average of 1 year
  The secondary objective is to demonstrate whether the aid of echo-assistance in the evaluation of the spine, performed by an experienced anesthesiologist, reduces the number of complications (particularly the number of attempts needed and the rate of dura puncture, (accidental dural puncture, ADP) in epidural catheter placement by inexperienced personnel (physicians in specialty training).
  The following outcomes will be considered to assess this objective:
  * number of traumatic punctures defined as: presence of redirects or number of punctures greater than one
  * median number of multiple punctures
  * number of women with failure (defined as number of punctures > 3)
  * number of accidental dural punctures (detected as CSF leaks).

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Guglielmetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy